CLINICAL TRIAL: NCT02629042
Title: Efficacy of Oral Prednisolone Versus Partial Endodontic Treatment on Pain Reduction in Emergency Care of Acute Irreversible Pulpitis of Mandibular Molars: Non Inferiority Randomized Clinical Trial
Brief Title: Efficacy of Oral Prednisolone on Pain Reduction in Emergency Care of Acute Irreversible Pulpitis
Acronym: PULPISOLONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2014/09
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Pulpitis
Keywords: Anesthesia; Corticosteroids; Dental Emergency; Irreversible Pulpitis; Mandibulae; Pain Management; Partial Endodontic Treatment
MeSH Terms: conditions — Pulpitis; Agnosia | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Procedure: Partial endodontic treatment under local and/or locoregional anesthesia
- Experimental (Experimental)
  Interventions: Drug: prednisolone

INTERVENTIONS:
Procedure: Partial endodontic treatment under local and/or locoregional anesthesia — The reference management consists in local and locoregional anesthesia of the molar and partial endodontic treatment. At the end of the emergency visit, all the patients, whatever their randomization group, will be given two types of antalgics and will be recommended to take them only if they have pain. Seventy-two hours after, all the patients, whatever their randomization will have endodontic treatment under local and locoregional anesthesia.
  Arms: Control
Drug: prednisolone — The evaluated intervention consists in per-os administration of prednisolone (1 mg / kg) during the emergency visit followed-up by one morning dose by day during three days. At the end of the emergency visit, all the patients, whatever their randomization group, will be given two types of antalgics and will be recommended to take them only if they have pain. Seventy-two hours after, all the patients, whatever their randomization will have endodontic treatment under local and locoregional anesthesia.
  Arms: Experimental

SUMMARY:
Irreversible pulpitis is an inflammatory condition of the dental pulp, highly painful, representing one of the main reasons for consulting dental emergency. The recommended emergency care is a partial endodontic treatment under local and/or locoregional anesthesia. The purpose of the emergency partial endodontic treatment is to stop the pain of pulpitis by removing a portion of the pulp. The final endodontic treatment is ideally performed 72 hours after. The literature reports major difficulty in obtaining adequate anesthesia in the mandible to perform partial endodontic treatment, especially for the mandibular molars. This results in a very painful care for the patient. The management of this type of emergency is costly in terms of equipment and time for health facilities. Patient comfort, cost saving and rationalization of the care time justify the search for an alternative to emergency partial endodontic treatment. In current practice, the short course oral corticotherapy is used in the management of oral pain from inflammatory origin. Glucocorticoids, thanks to their anti-inflammatory action, can neutralize the inflammatory mediators and thus pain. The pulp inflammation can be treated with this molecule: the effectiveness of intraosseous local steroid injection for irreversible pulpitis of mandibular molars has already been shown but results in local comorbidities and requires specific device. Oral administration of short-course prednisolone is simple and safe but its effectiveness to manage pain caused by irreversible pulpitis has not yet been demonstrated. Per-os administration of prednisolone has a very high (90%) and rapid (≤ 4 hours) bioavailability. No difference in effectiveness between intravenous and oral administration of this molecule was reported. This oral treatment could limit comorbidities and technical difficulties related to intraosseous injection and could delay the endodontic treatment to 72 hours in optimal conditions of anesthesia for the patient. Despite the difficulties described for the partial endodontic treatment, it is very effective in pain reduction and can reach 100% of success. Therefore a non-inferiority design was chosen to compare the effect of a short-course oral corticotherapy to a partial endodontic treatment for the reduction of pain at the emergency care of the irreversible pulpitis in mandibular molars. The intervention arm will receive an oral dose of prednisolone (1 mg/kg) during the emergency visit followed-up by one morning dose by day during three days and the reference arm will have partial endodontic treatment. Both groups will have planned complete endodontic treatment 72 hours after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of irreversible pulpitis on a mandibular molar,
* ASA1 or ASA2 score (American Society of Anesthesiologists)
* Age between 18 and 70 years (of either gender)
* Ability to give written informed consent
* Affiliation to a health insurance scheme
* Agreement to be contacted by phone 24h after the emergency visit
* Availability to come back 72 hours after the emergency visit for endodontic treatment

Exclusion Criteria:

* Diagnosis of reversible pulpitis, acute apical periodontitis, periodontal lesion of endodontic origin or dentin syndrome
* Not retainable tooth requiring extraction
* Contraindication of endodontic treatment (endocarditis risk) or local anaesthesia
* Contraindication for the prescription of glucocorticoids, paracetamol or codeine,
* Oral infection, viral disease in evolution (hepatitis, herpes zoster, .. ),
* Machine operators ,
* Psychosis uncontrolled by treatment, or chronic consumption of drugs or alcohol
* Allergy to one or more of the components,
* Diabetes, drug intake with direct interaction with glucocorticoids, paracetamol or codeine,
* Woman of child-bearing age without contraceptive, pregnancy, breastfeeding
* Not able to give informed consent,
* Participating in another interventional study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity on a numeric scale | 24 hours after the emergency visit (inclusion)

SECONDARY OUTCOMES:
The number of antalgic drugs taken after the emergency visit | 72 hours after the emergency visit (inclusion)
The number of patients coming back to consultation at 72h | 72 hours after the emergency visit (inclusion)
The number of injected anesthetic cartridges when performing the endodontic treatment | 72 hours after the emergency visit (inclusion)
Patient's comfort evaluation during the endodontic treatment using a questionnaire with numeric scales | 72 hours after the emergency visit (inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Elise ARRIVE, Study Chair — USMR, CHU de Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Kerouredan O, Jallon L, Perez P, Germain C, Peli JF, Oriez D, Fricain JC, Arrive E, Devillard R. Efficacy of orally administered prednisolone versus partial endodontic treatment on pain reduction in emergency care of acute irreversible pulpitis of mandibular molars: study protocol for a randomized controlled trial. Trials. 2017 Mar 28;18(1):141. doi: 10.1186/s13063-017-1883-x. PMID 28351379